CLINICAL TRIAL: NCT06247059
Title: Reducing Respiratory Virus Transmission in Bangladeshi Classrooms
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Principal Investigator, Stephen P Luby, Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 73657
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: SARS-CoV2 Infection; Influenza Viral Infections; Respiratory Viral Infection
Keywords: Bangladesh; Indoor air quality; Air cleaning; Respiratory viral infections; Influenza; SARS-CoV2; Air filtration; Ultraviolet germicidal irradiation; Global health
MeSH Terms: conditions — COVID-19; Influenza, Human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Box Fan (Experimental): Classrooms receive box fans equipped with a filter.
  Interventions: Device: Box Fan
- UV Germicidal Irradiation Lamp Unit (Experimental): Classrooms receive UV germicidal irradiation lamp unit(s).
  Interventions: Device: UV Germicidal Irradiation Lamp Unit
- Combined: Box Fan and UV Germicidal Irradiation Lamp Units (Experimental): Classrooms receive box fans equipped with a filter and UV germicidal irradiation lamp unit(s).
  Interventions: Device: Combined: Box Fan and UV Germicidal Irradiation Lamp Units
- Non-Interventional Control (No Intervention): Classrooms receive no intervention to their standard classroom setup.

INTERVENTIONS:
Device: Box Fan — Classrooms assigned to this arm will be equipped with 2 - 8 box fans each with a single minimum efficiency reporting value-14 (MERV-14) filter sufficient to increase effective air changes per hour to 12 based on the clean air delivery rate measured in cubic feet per minute of the box fan + filter * 60 divided by the room volume.
  Arms: Box Fan
Device: UV Germicidal Irradiation Lamp Unit — Classrooms assigned to this arm will be equipped with one or two 222nm wavelength light ultraviolet germicidal irradiation lamp units (number of units per classroom based on room volume).
  Arms: UV Germicidal Irradiation Lamp Unit
Device: Combined: Box Fan and UV Germicidal Irradiation Lamp Units — Classrooms assigned to this arm will be equipped with both box fans and UV germicidal irradiation lamp units.
  Arms: Combined: Box Fan and UV Germicidal Irradiation Lamp Units

SUMMARY:
This study will test if affordable air cleaning devices (box fans with a filter attached and/or ultraviolet light lamps) installed in classrooms can reduce the number of viral respiratory illnesses schoolchildren experience.

DETAILED DESCRIPTION:
This cluster-randomized controlled trial in Bangladesh schools will examine whether low-cost air filtration and/or human-safe ultraviolet germicidal light interventions can reduce the incidence of schoolchildren's respiratory viral infections. The main study objectives are:

1. Pilot and optimize an intervention to filter classroom air.
2. Pilot and optimize an intervention to treat classroom air with ultraviolet light.
3. Assess the separate and combined effect of air filtration and ultraviolet light on the incidence of polymerase chain reaction (PCR) confirmed illness from respiratory viruses.

Methods: The study will take place in 60 government primary schools in Dhaka, Bangladesh. Within each enrolled school, 5 classrooms of students in grades 3, 4 and 5 will be randomly assigned to receive:

1. Box fans with a filter attachment.
2. 220 nanometer (nm) wavelength ultraviolet light air cleaner lamps.
3. Both the box fans with a filter and the 220 nm ultraviolet lamps.
4. No device: a control group that receives no additional device ("standard of care"). Two classrooms within each school will be assigned as controls.

Why does this matter?: Clarifying the impact of low-cost practical solutions could support the adoption of these strategies that could reduce influenza and severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) transmission in schools in order to reduce the burden of respiratory illness in these communities.

ELIGIBILITY:
Inclusion Criteria:

* Schoolchildren of Bangladesh Government-run primary schools in Dhaka, Bangladesh ages 9 - 12 years, of all gender identifiers (male, female, transgender, prefer not to designate), without specific ethnic selection amongst standard school children of Bangladesh government schools in Dhaka, Bangladesh.

Exclusion Criteria:

* School children of non-Bangladesh Government-run primary schools and/or schoolchildren who do not attend a Bangladesh Government-run primary school in Dhaka, Bangladesh.
* School children who are not able to or have a contraindication with the ability to comply with study procedures.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20000 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Total number of symptomatic respiratory illness episodes due to either Influenza or SARS- CoV-2 | Over 40 weeks of observation
  Study personnel will visit each school twice weekly. They will identify any students within the study classrooms who were absent or who have symptoms consistent with the World Health Organization (WHO) definition of influenza like illness. For children who were absent or who have symptoms, study personnel will visit the child's home, and if the student's parent provides informed consent, collect more detailed information on signs and symptoms, and a throat swab from the child. The throat swab will be placed on viral transport media, placed on ice and transported to the One Health Laboratory at the International Centre for Diarrhoeal Disease Research, Bangladesh (icddr,b). One aliquot from the specimen will be analyzed for Influenza A, Influenza B, and SARS-CoV-2. In the laboratory, nucleic acid in the throat swab specimen will be extracted and one-step real-time (RT)-PCR conducted to assess the presence of RNA from Influenza A, Influenza B or SARS-CoV-2.

SECONDARY OUTCOMES:
Total number of symptomatic influenza-like illness episodes | Over 40 weeks of observation
  Study personnel will visit each school twice weekly. They will identify any students within the study classrooms who were absent or who have symptoms consistent with the WHO definition of influenza like illness.
Total number of symptomatic influenza episodes | Over 40 weeks of observation
  Study personnel will visit each school twice weekly. They will identify any students within the study classrooms who were absent or who have symptoms consistent with the WHO definition of influenza like illness. For children who were absent or who have symptoms, study personnel will visit the child's home, and if the student's parent provides informed consent, collect more detailed information on signs and symptoms, and a throat swab from the child. The throat swab will be placed on viral transport media, placed on ice and transported to the One Health Laboratory at icddr,b. One aliquot from the specimen will be analyzed for Influenza A or Influenza B. In the laboratory, nucleic acid in the throat swab specimen will be extracted and one-step real-time RT-PCR conducted to assess the presence of RNA from Influenza A or Influenza B.
Total number of symptomatic SARS-CoV2 episodes | Over 40 weeks of observation
  Study personnel will visit each school twice weekly. They will identify any students within the study classrooms who were absent or who have symptoms consistent with the WHO definition of influenza like illness. For children who were absent or who have symptoms, study personnel will visit the child's home, and if the student's parent provides informed consent, collect more detailed information on signs and symptoms, and a throat swab from the child. The throat swab will be placed on viral transport media, placed on ice and transported to the One Health Laboratory at icddr,b. One aliquot from the specimen will be analyzed for SARS-CoV2. In the laboratory, nucleic acid in the throat swab specimen will be extracted and one-step real-time RT-PCR conducted to assess the presence of RNA from SARS-CoV2.
Total number of student absentee episodes | Over 40 weeks of observation
  Study personnel will visit each school twice weekly. They will identify any students within the study classrooms who were absent.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen P Luby, MD, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No